CLINICAL TRIAL: NCT07330921
Title: Development and Effectiveness of the Participatory Adapted 3D Seating System (SSAP3D) and Its Impact on the Daily Performance of Children With Neuromotor Dysfunction and Their Families: Pilot Study
Brief Title: Development and Effectiveness of the Participatory Adapted 3D Sedentation System (SSAP3D).
Acronym: SSAP3D
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Collaborators: Universidad Pontificia Comillas (Other)
Responsible Party: Principal Investigator, Sandra Calvo Carrión, Phd, Instituto de Investigación Sanitaria Aragón
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UZ-Asientos 3D
Record Dates: First submitted 2025-09-22; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Neuromotor Dysfunction
Keywords: Performance; Children; Seating System; 3D Technology; Quality of Life

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SSAP3D Intervention (Experimental): Participants will use the SSAP3D during the whole day by the child and the family for 6 weeks.
  At the beginning of the study, will carry out a session for taking body measurements and collecting data through the scanning of the participant.
  From this data collection, the SSAP3D will be digitally created. After all the necessary modifications have been made, the seat will be printed using FDM 3D Printer. Once the printing is finished, the removable systems and padding will be adjusted and placed by the designed interlocking systems.
  Three weeks after the data collection session, the SSAP3D will be delivered to the family and the 6-weeks intervention will begin.
  The correct elaboration of the device will be checked. Also, basic guidelines on the correct use of the seat, moments of use and maintenance of the seat will be explained to both the child and the families. This information will also be communicated to the school staff and to the different early care centers they attend.
  Interventions: Device: SSAP3D Intervention

INTERVENTIONS:
Device: SSAP3D Intervention — The intervention is the same for the whole sample but with deferent sequences: group 1 will perform the intervention following the sequence "SSAP3D + conventional system" and group 2 will perform the intervention with the opposite sequence, "conventional system + SSAP3D". Both groups will use 6 weeks the SSAP3D and 6 weeks the conventional system.
  During the 6 weeks of intervention using SSAP3D, 2 online follow-up sessions will be carried out with the family (weeks 6 and 8 for group 1; weeks 9 and 11 for group 2) with the aim of supervising the correct use and maintenance of the seat, as well as resolving possible doubts and/or the need to make anu modifications or adjustments to the seat, both in the family and school environment of the participant.

SUMMARY:
Problems with postural control cause difficulties in children's motor development, leading to significant structural and functional complications, including pelvic obliquity, scoliosis, and asymmetries in both active and passive ranges of motion. All these difficulties affecting posture control have a negative impact on children's functional autonomy and independent participation in their daily activities, as well as on their interaction with different environments, mainly family, social, and educational. In view of this situation, the 3D Adaptive Sitting System "SSAP3D", a 3D pelvic ser with a self-extracting abductor cushion, is proposed as an alternative.

The main objective is to develop and test a novel 3D-printed adaptive seating system, called SSAP3D, tailored to individual needs of children with Neuromotor Dysfunction, to assess whether it promotes the functional performance of children in their daily and meaningful activities.

A secondary objective is to analyze whether the use of SSAP3D promotes the children's participation in different environments compared to a conventional seated system.

The sample is estimated at 12 children, all of them were between 2-6 years old and with Neuromotor Dysfunction from early attention centers, as well as from private rehabilitation centers or associations.

The intervention program will be the same for each participant, but in different temporal order. 6 children will use during the first 6 weeks the 3D seat and the following 6 weeks their usual seating system; the others 6 children inverted order. The 3D seat will be made individually for each child. The device will be delivered 3 weeks after the scanning-data collection accompanied by guidelines for use. There will be 2 online follow-up sessions.

Hypothesis: the implementation of the SSAP3D allows to ensure the postural requirements of children with Neuromotor Dysfunction and to favor their functional performance in daily and meaningful activities at home, at school and in their community. In addition, it will have a positive impact on the quality of life perceived by the families related to the characteristics of the seat.

DETAILED DESCRIPTION:
This project employs a pilot study of a crossover clinical trial with two groups with two deferent sequences: group 1 will perform the intervention following the sequence SSAP3D + conventional system and group 2 will perform the intervention with the opposite sequence, conventional system + SSAP3D.

Intervention Protocol:

At the beginning of the study, both groups will carry out a 30-minute evaluation session for taking body measurements and collecting data through the scanning of the participant.

Through these measures, the investigators will design a SSAP3D for the participant, an individual 3D printed seat. Three weeks after the data collection session, the SSAP3D will be delivered to the family with a basic guideline on the correct use of the seat.

The intervention, which consist in the use of the SSAP3D during the whole day by the child and the family for 6 weeks, will be controlled by two online follow-up sessions with the family.

Quantitative Data Collection Protocol:

The quantitative assessment will be carried out by two physiotherapists previously trained in the selected measurement tools and with extensive clinical experience in the field of neurorehabilitation. There will be an evaluation site, located at the facilities of the "Asociacion para la Investigación en Discapacidad Motriz" (AIDIMO), in Zaragoza. The evaluations will last approximately 90 minutes. The study will have 4 evaluation times: E1: assessment prior to the start of the study; E2: post-intervention assessment (SSAP3D in the case of group 1 and usual seated system in the case of group 2); E3: post-intervention assessment (usual seated system in the case of group 1 and SSAP3D in the case of group 2); ES1: follow-up assessment 3 months after the end of the study. Outcome measurement tolls 2 and 2 will be videotaped with audio for better analysis by the evaluators, and, in case of any doubt, to be able of consult this material to corroborate the results.

Data Analysis Approach:

Quantitative data will be analyzed using the statical program IBM SPSS Statics Version 29.0 (SPSS Inc., Chicago, Illinois, USA). The normality of distribution of quantitative variables will be verified using the Shapiro-Wilk test, which is suitable for small samples and provides an accurate assessment of normality, Descriptive statics will be presented as mean ± standard deviation or median [interquartile range] for continuous parameters, and as frequency (%) for categorical data. Baseline measurements will be compared between groups using Student's t-test for independent samples, the Mann-Whitney U test, and the chi-square test, as appropriate for the nature of the variable. An intergroup (between groups) and intragroup (within each group) analysis will be performed using a mixed model analysis of variance (ANOVA) one-way and for repeated measures with Bonferroni pairwise post hoc comparisons that adjusts the significance level for multiple comparisons. In case the distribution is not normal. A nonparametric analysis will be performed using the Mann-Whitney U test to compare at the intergroup level and Friedman's test with Tukey's post hoc test to identify differences at the intragroup level. In addition, effect size will be calculated using Cohen's d coefficient, which is interpreted as small (d=0.2), medium (d=0.5) or large (d>0.8). The significance level will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Medical Situation of Neuromotor Disfunction
* Be user of some type of adapted seating system
* Age between 2-6 years
* Have head control levels of 3 to 8 on the Level of Sitting Scale (LSS)
* Be able to maintain a standing position for at least 10 seconds, with or without external assistance.

Exclusion Criteria:

* Presenting moderate or severe cognitive impairment, which generates significant difficulties in understanding the instructions given by the evaluator
* Having suffered a traumatic injury o surgical process in the 6 months prior to the start of the study or during the study

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2025-12-13 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Performance | from enrollment to the end of intervention, as in the two-follow-up assessment, assessed up to 9 months
  Change in the score on the Pediatric Evaluation of Disability Inventory-Computer Adaptive Test (PEDI-CAT). The PEDI-CAT is a computerized and adaptive questionnaire completed by the family that measures the child's functional performance in the areas of activities of daily life, mobility, social/cognitive function and responsibility in complex daily tasks. In addition, in children with Neuromotor Dysfunction, the PEDI-CAT has been shown to be a valid instrument to measure functional ability.
  30-70: Considered the expected range for age, indicating normal functional capacity.
  < 30: Suggests lower than expected functional capacity for age.

SECONDARY OUTCOMES:
Postural control | from enrollment to the end of intervention, as in the two-follow-up assessment, assessed up to 9 months
  Changes in the score of Postural control measure (SPCM): a 34-item scale designed to measure changes in postural alignment and functional movement produced by an intervention focused on adapted seating systems. It has shown good psychometric properties for children with Neuromotor Dysfunction.
  1. Postural Alignment Section (SPCM-A): 22 items, scored on a 4-point ordinal scale. From 1: Neutral alignment (typical posture), to 4: Severe deviation
  2. Functional Movement Section (SPCM-F): 12 items, scored on a 4-point ordinal scale. From 1: Unable to initiate the task, to 4: Successful completion of the task
Functionality of upper extremity | from enrollment to the end of intervention, as in the two-follow-up assessment, assessed up to 9 months
  Change in the score on the Box and Block Test (BBT). The BBT measures the functionality of the upper extremity in children with Neuromotor Dysfunction, specifically gross motor dexterity in a unimanual way in terms of speed and accuracy.
Achievement of Functional goals | from enrollment to the end of intervention, as in the two-follow-up assessment, assessed up to 9 months
  Change in the score on the Canadian Occupational Performance Measure (COPM). The COPM is designed to identify occupational performance problems through a semi-structured, clinically useful and responsive interview that allows for person-centered practice. The COPM will be used to establish three occupational performance problems in each child, which will be identified by the family and used as functional treatment goals.
  * Importance Score: The client rates the importance of each activity identified for their life, using an ordinal scale from 1 to 10.
    1: Not important at all. 10: Extremely important.
  * Performance: How well do you currently perform the activity?
    1: Unable to perform at all (or with great difficulty). 10: Able to perform extremely well (or without difficulty).
  * Satisfaction: How satisfied are you with your current level of performance in this activity? 1: Not at all satisfied. 10: Extremely satisfied.
Participation in different environments | from enrollment to the end of intervention, as in the two-follow-up assessment, assessed up to 9 months
  Change in the score on the Young Children's Participation and Environment Measure (YC-PEM). Measurement instrument filled out by the parents or primary caregiver, which analyzes the different activities of the child between 0-5.9 years of age, assessing their level of participation and the qualities of the environment in which they develop.
  1. Frequency of Participation 8 points, from 0 (never) to 7 (one or more times a day). A higher score indicates greater frequency of participation in these activities.
  2. Level of Involvement 5 points, from 1 (not very envolved) to 5 (Very involved.).A higher score indicates a greater level of interaction and active participation in activities.
  3. Percentage of Desired Change Percentage (0% to 100%). A lower percentage suggests greater satisfaction with the child's current participation.
     A higher percentage indicates that the caregiver desires change.
  4. Environmental Support (Facilitators and Barriers) Percentage (0% to 100%)
Quality of Life | from enrollment to the end of intervention, as in the two-follow-up assessment, assessed up to 9 months
  Change in the score on the Pediatric Quality of Life Inventory (PedsQL): a tool for measuring health-related quality of life in children and adolescents aged 2 to 18, assessing physical, emotional, social, and school functioning. In the versions for younger children, a report completed by parents is used. Widely adapted and validated in Spanish.
  * Ages 5-7 (Parent-report): 3-point scale.
  * Ages 2-4 (Parent report): 3-point scale.
  To calculate the final scores, the items are reversed and linearly transformed to a scale of 0 to 100, where:
  * 0 (frequent problem) becomes 0 (low HRQoL).
  * 4 (never a problem) becomes 100 (high HRQoL) High Scores (close to 100): Indicate excellent quality of life and few health problems.
  Low Scores (close to 0): Indicate poor quality of life and significant health problems.
Family Satisfaction | from enrollment to the end of intervention, as in the two-follow-up assessment, assessed up to 9 months
  Change in the score on the Family Impact of Assistive Technology for Adapting Sitting (FIAT-AS). It is a questionnaire completed by parents that measures the functional status and change in habits of the child with Neuromotor Dysfunction and the family as influenced by interventions focused on adapted seating systems.
  Parents respond to 64 items (originally 89) using a 7-point Likert scale, ranging from:
  1: Strongly Disagree 7: Strongly Agree. High Scores (close to 7): Indicate a positive impact and better functioning of the child and family in that specific dimension. For example, a high score on "Autonomy" means that the child is perceived as very autonomous.
  Low scores (close to 1): Indicate a negative impact, poorer functioning, or the presence of significant barriers. For example, a low score on "Caregiver Relief" means that the caregiver experiences little relief from their tasks.
Postural control | from enrollment to the end of intervention, as in the two-follow-up assessment, assessed up to 9 months
  Changes in the score of Segmental assessment of trunk control (SATCo): validated and reliable scale for children with Neuromotor Dysfunction and for neuromotor disorders, which measures the degree of trunk control its different segments while seated.
  The score is based on a "pass/fail" (present/absent) system for control in each segment, under three specific conditions at each level:
  Static Control Active (Anticipatory) Control Reactive Control
  For data analysis and clinical follow-up, an ordinal numerical value is assigned to each level of control achieved:
  1. Functional control of the head only (the trunk is unstable and requires maximum support).
  2. Control of the head and upper cervical segments.
  3. Control of the head and upper chest.
  4. Control of the head and most of the thorax.
  5. Control of the head, thorax, and upper abdomen.
  6. Control of the entire spine except the pelvis
  7. Complete trunk control, no manual support required

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Calvo, PhD, Principal Investigator — Universidad de Zaragoza
Locations (1):
- AIDIMO (Asociación para la Investigación en la Discapacidad Motriz), Zaragoza, Zaragoza, Spain